CLINICAL TRIAL: NCT04790292
Title: Impact of Dexamethasone Added to Intra-articular Morphine and Bupivacaine for Post-operative Analgesia After Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba Fouad Abd El-Aziz Toulan, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU MS 20/2020
Record Dates: First submitted 2021-03-01; First posted 2021-03-10 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia
Keywords: Dexamethasone; Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group M (Active Comparator): group M 10mg morphine +0.25% bupivacaine
  Interventions: Drug: group M
- group MD (Active Comparator): group MD 10mg morphine + 8mg dexamethasone +0.25% bupivacaine
  Interventions: Drug: group MD

INTERVENTIONS:
Drug: group M — 10mg morphine in 5ml normal saline + 10ml of 0.25% bupivacaine ( total volume 15 ml) were injected intra-articularly
  Arms: group M
Drug: group MD — 10mg morphine + 8mg dexamethasone completed to 5 ml with normal saline + 10 ml of 0.25% bupivacaine (total volume of 15ml) were injected intra-articularly
  Arms: group MD

SUMMARY:
A randomized double-blinded clinical trial was carried out on 40 patients undergoing knee arthroscopy. Patients were divided randomly into two equal groups. All drugs used were injected intra-articularly at the end of arthroscopy. In the control group, patients were administered 10mg morphine added to bupivacaine 25mg. In the study group, patients were administered 10mg morphine and 8mg dexamethasone added to bupivacaine 25mg. Visual analog score for pain at rest and movement, time to first analgesic request, total analgesic consumption, duration of analgesia and adverse effects were recorded.

ELIGIBILITY:
Minimum Age: 18 years Maximum Age: 65 years Sex: Both Gender Based: No Accepts Healthy Volunteers: No

Criteria:

Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* Scheduled for minor arthroscopic knee surgeries (meniscectomy, chondroplasty, minor ligament repair and diagnostic arthroscopy)

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status above (II)
* Undergoing major knee surgeries
* History of allergies to any of the used drugs
* History of diabetes mellitus
* Contraindications of morphine use (e.g. asthmatic patient, chronic obstructive pulmonary disease, and addiction)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
visual analogue score(VAS) at rest and movement | first 24 hours post operative
  visual analogue score(VAS) will be used to measure pain score (VAS score 0 cm= no pain, VAS score 10 cm = worst possible pain) when the patient is fully conscious (0) and at 2, 4, 6, 8, 10, 12, 18, 24 hours post-operatively

SECONDARY OUTCOMES:
Rescue analgesia time | first 24 hours post operative
  Time to first analgesia requirement (considering the extubation is zero time)
Total analgesic consumption | first 24 hours post operative
  intramuscular diclofenac sodium 75mg will be given as rescue analgesic when VAS ≥ 4. Total diclofenac consumption will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Heba F Abd El-Aziz Toulan, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No